CLINICAL TRIAL: NCT04083001
Title: An Open, Multi-centre Study to Assess the Safety and Tolerability of RGTA® (OTR4132) in Patients With Acute Ischemic Stroke (AIS)
Brief Title: An Open, Study to Assess the Safety of RGTA® (OTR4132) in Patients With Acute Ischemic Stroke (AIS)
Acronym: MATRISS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Organ, Tissue, Regeneration, Repair and Replacement (Industry)
Collaborators: European Commission (Other); Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A03117-48
Record Dates: First submitted 2019-09-03; First posted 2019-09-10 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Stroke, Acute
Keywords: Stroke; FIM; OTR3
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: open study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OTR4132MD (Experimental): One medical device will be administrated as a one shot-dose to the patient. The respective total dose of OTR4132 received by a patient will be one of the following: 0,20 mg, 0,50 mg, 1 mg, 1,5 mg, 2 mg and 2,5 mg.
  Interventions: Device: OTR4132MD

INTERVENTIONS:
Device: OTR4132MD — According to Regulation (EU) 2017/745(MDR), OTR4132-MD is an implantable medical device, for short term use which is specifically intended for use in direct contact with systemic circulation system.
  OTR4132-MD is by definition intended to come into contact with the patient when being injected. It is administered through intra-arterial injection, in an one-shot dose and the majority of the product is eliminated within 24 hours.

SUMMARY:
RGTA® (ReGeneraTing Agent) are synthetic polysaccharides mimicking extra-cellular matrix scaffold elements and protective agents called Heparan Sulphates (HSPGs).

OTR4132-MD is provided as a sterile injectable medical device. OTR4132-MD is indicated in anterior circulation acute ischemic stroke (AIS) patients re-vascularized (TICI score 2b - 3) by endovascular thrombectomy combined or not with thrombolysis.

DETAILED DESCRIPTION:
The promising results of OTR4132-MD in the treatment of acute ischemic stroke in animal studies and the excellent results of biocompatibility tests reported in the Investigator's Brochure allowed to design a clinical investigation in humans named MATRISS. As this is a First-In-Man (FIM) study assessing OTR4132-MD, it is designed as a single ascending dose (SAD) to evaluate the safety, tolerability of a single intra-arterial injection of OTR4132-MD in AIS patients treated with thrombectomy combined or not with thrombolysis.

The FIM will include up to 19 patients in up to six dose groups. Each group will comprise 3 subjects. This FIM study will also monitor a dose response relationship in humans: lesion volume change throughout the study period. Patients will be given a single intra-arterial injection of OTR4132-MD with a predefined dose of OTR4132. In the first dose group, the OTR4132 dose is 0.20 mg.

The results of this study will serve as a groundwork for the design of a pivotal study in the intended patient population.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients for this study will be included if all of the following conditions are met:

1. Age between 45 and 80 years
2. Acute ischemic stroke in anterior circulation territory, identified by magnetic resonance imaging (MRI)
3. Occlusion of anterior circulation i.e. internal carotid artery (ICA) or proximal middle cerebral artery (MCA) (M1 and/or M2 segment)
4. Volume of the infarcted lesion estimated below two thirds of the MCA territory (diffusion MRI sequence)
5. Endovascular thrombectomy initiated within 6 hours of stroke onset with known stroke onset time or Endovascular thrombectomy initiated within 6 to 16 hours of symptoms onset (last know well in case of unwitnessed onset) with a mismatch on brain MRI defined in *.
6. Recanalization confirmed by angiography after endovascular treatment: TICI grade 2b - 3
7. NIHSS at pre-screening (National Institute of Health Stroke Scale/Score), including hand testing: between 11 and 25
8. No significant pre-stroke disability (pre-stroke modified Rankin Score (mRS): 0-1
9. Able to follow neuro-rehabilitation programme
10. Patient** or legally authorized representative (family member or trusted person if patient unable to give consent) or independent physician (if patient unable to give consent and if an authorized representative cannot be reached) has signed informed consent).

    * Perfusion core/penumbra mismatch:

      * Infarct core volume <70 mL
      * and critically hypoperfused volume/infarct core volume >1.8
      * and mismatch volume >15mL ** Patients unable to give consent at baseline will go through a deferred consent procedure to continue the study

Exclusion Criteria:

* Eligible patients for this study will not be included if any of the following conditions are present:

  1. Previous symptomatic stroke
  2. Pre-existing medical, neurological, or psychiatric disease that would confound the neurological evaluation
  3. Contra-indication to MRI
  4. Evidence of intracranial haemorrhage (ICH)
  5. At the discretion of the investigator, patients with co-morbidities associated with a life expectancy of less than 3 months or co-morbidities that could influence the study results or would complicate assessment of outcomes (e.g. dementia, psychiatric disease) or would make clinical follow-up difficult
  6. History of allergy or anaphylactic reactions to any of the ingredients of OTR4132-MD or heparinoids
  7. History of Hypersensitivity or anaphylactic reactions to iodinated contrast media
  8. Severe renal failure with glomerular filtration rate (GFR) < 30 mL/min
  9. Severe uncontrolled arterial hypertension e.g. systolic blood pressure > 185 mmHg or diastolic blood pressure > 110 mmHg, or intravenous medication necessary to reduce blood pressure
  10. Increased risk of haemorrhage (such as medical history of significant bleeding disorders, major surgery or significant trauma in the past 3 months, any history of central nervous damage or suspected intracranial haemorrhage, symptoms suggestive of subarachnoid haemorrhage, even if the MRI is normal, international normalized ratio (INR)>1.3 or activated partial thromboplastin time (aPTT)>ULN (upper limit of normal)
  11. Suspected cerebral vasculitis based on medical history and imaging
  12. Occlusions in multiple vascular territories
  13. Evidence of intracranial tumour
  14. Evidence of any prior intracranial intervention (i.e. neurosurgery, endovascular intervention)
  15. Worsening of medical or neurological conditions or per-procedures complications
  16. Any other serious, advanced, or terminal illness (investigator judgment)
  17. Pregnant or breastfeeding or women without an adequate contraceptive method
  18. Current participation in another investigation drug or device study
  19. The patient is not a member or beneficiary of the French social security system

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Rate of severe adverse events device related and dose limiting | 7 Days
  Severe adverse events

SECONDARY OUTCOMES:
Survival rates | 24 hours, 7 Days, 30 Days, 90 Days
  survival rates
All cause death | 24 hours, 7 Days, 30 Days, 90 Days
  All cause death
Stroke related death | 24 hours, 7 Days, 30 Days, 90 Days
  Stroke related death
Rate of device related adverse events (AEs) and serious adverse events (SAEs) | 24 hours, 7 Days, 30 Days, 90 Days
  rate of device related adverse events
Rate of adverse events (AEs) and serious adverse events (SAEs) procedure related | 24 hours, 7 Days, 30 Days, 90 Days
  Rate of AEs and SAEs propcedure related
Symptomatic intracranial haemorrhage | 24 hours, 7 Days, 30 Days, 90 Days
  Intracranial haemorrhage
Brain oedema on 24-hour follow-up imaging | 24 hours
  brain oedema
New ischaemic lesions | 24 hours
  Ischaemic lesions in new territories on 24-hours follow-up imaging

OTHER OUTCOMES:
Revascularization on 24-hour follow-up imaging | 24 Hours
  Revascularization on 24-hour follow-up imaging

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Detante, Principal Investigator — CHU Grenoble Alpes
Locations (3):
- France (3):
  - CHU Grenoble Alpes, Grenoble, Auvergne-Rhône-Alpes
  - CHU Nancy, Nancy, Grand Est
  - CHU Bordeaux Pellegrin, Bordeaux, Nouvelle-Aquitaine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barreau X, Anxionnat R, Heck O, Sibon I, Rosso C, Oppenheim C, Moniche F, Sedel F, Chiappini F, Choppin A, Inizan M, Barritault D, Detante O. Intra-arterial Injection of OTR4132, a Novel Neuroprotector in Acute Ischemic Stroke: The MaTRISS Trial. Clin Drug Investig. 2025 Nov;45(11):877-887. doi: 10.1007/s40261-025-01487-y. Epub 2025 Oct 2. PMID 41037228